CLINICAL TRIAL: NCT07212855
Title: Analysis of the Effectiveness of the Use of Glycine Powder and an Angled Implant Brush in Oral Hygiene Procedures in Patients Rehabilitated With Columbus Bridge Protocol: a Factorial Randomized Study
Brief Title: Use of Glycine Powder and an Angled Implant Brush in Oral Hygiene Procedures in Patients Rehabilitated With Columbus Bridge Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Jacopo Lanzetti, Doctor in Dental Hygiene, University of Turin, Italy
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 134/2023
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Full Arch Fixed Prosthesis
Keywords: professional oral hygiene; domiciliary oral hygiene; full arch fixed prosthesis; implant disease prevention

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- professional oral hygiene with glycine and domiciliary oral hygiene with angle toothbrush (Experimental): Patients randomized to the Test group for professional oral hygiene underwent professional removal of hard and soft deposits using titanium curettes, spongy interdental floss, and air-polishing with glycine powder. The glycine powder used had a particle size of 25 μm and was applied using a supragingival nozzle positioned 3 mm from the prosthetic restoration, with particular attention given to the areas in direct contact with the mucosa.
  Patients randomized to the Test group for domiciliary oral hygiene procedures - were motivated and instructed to use an angled-handle toothbrush (Specialist Implant, Curasept S.p.A., Saronno, Italy), in addition to a standard toothbrush and implant floss. The specific design of the angled handle was intended to facilitate access to areas that are difficult to clean. In patients rehabilitated with full-arch implant-supported prostheses, these areas typically include distal cantilevers and surfaces in direct contact with the mucosa.
  Interventions: Procedure: Professional oral hygiene with glycine powder; Device: Domiciliary oral hygiene with angle toothbrush
- professional oral hygiene with glycine and domiciliary oral hygiene with standard toothbrush (Active Comparator): Patients randomized to the Test group for professional oral hygiene underwent professional removal of hard and soft deposits using titanium curettes, spongy interdental floss, and air-polishing with glycine powder. The glycine powder used had a particle size of 25 μm and was applied using a supragingival nozzle positioned 3 mm from the prosthetic restoration, with particular attention given to the areas in direct contact with the mucosa.
  Patients randomized to the Control group for domiciliary oral hygiene procedures were motivated exclusively to use a standard toothbrush and implant floss.
  Interventions: Procedure: Professional oral hygiene with glycine powder
- professional oral hygiene without glycine and domiciliary oral hygiene with angle toothbrush (Active Comparator): Patients randomized to the Control group for professional oral hygiene underwent professional removal of hard and soft deposits exclusively by means of titanium curettes and spongy interdental floss.
  Patients randomized to the Test group for domiciliary oral hygiene procedures - were motivated and instructed to use an angled-handle toothbrush (Specialist Implant, Curasept S.p.A., Saronno, Italy), in addition to a standard toothbrush and implant floss. The specific design of the angled handle was intended to facilitate access to areas that are difficult to clean. In patients rehabilitated with full-arch implant-supported prostheses, these areas typically include distal cantilevers and surfaces in direct contact with the mucosa.
  Interventions: Device: Domiciliary oral hygiene with angle toothbrush
- professional oral hygiene without glycine and domiciliary oral hygiene with standard toothbrush (No Intervention): Patients randomized to the Control group for professional oral hygiene underwent professional removal of hard and soft deposits exclusively by means of titanium curettes and spongy interdental floss.
  Patients randomized to the Control group for domiciliary oral hygiene procedures were motivated exclusively to use a standard toothbrush and implant floss.

INTERVENTIONS:
Procedure: Professional oral hygiene with glycine powder — Professional removal of hard and soft deposits using titanium curettes, spongy interdental floss, and air-polishing with glycine powder. The glycine powder used had a particle size of 25 μm and was applied using a supragingival nozzle positioned 3 mm from the prosthetic restoration, with particular attention given to the areas in direct contact with the mucosa.
  Arms: professional oral hygiene with glycine and domiciliary oral hygiene with angle toothbrush; professional oral hygiene with glycine and domiciliary oral hygiene with standard toothbrush
Device: Domiciliary oral hygiene with angle toothbrush — Patients were motivated and instructed to use an angled-handle toothbrush (Specialist Implant, Curasept S.p.A., Saronno, Italy), in addition to a standard toothbrush and implant floss. The specific design of the angled handle was intended to facilitate access to areas that are difficult to clean. In patients rehabilitated with full-arch implant-supported prostheses, these areas typically include distal cantilevers and surfaces in direct contact with the mucosa.
  Arms: professional oral hygiene with glycine and domiciliary oral hygiene with angle toothbrush; professional oral hygiene without glycine and domiciliary oral hygiene with angle toothbrush

SUMMARY:
Dental implants are widely employed in modern dentistry for the rehabilitation of patients affected by edentulism, whether limited to a single missing tooth, multiple adjacent teeth, or involving complete dental arches. In particular, full-arch rehabilitations provide both functional and aesthetic restoration of completely edentulous arches or of severely compromised dentitions that the preservation of the remaining teeth is no longer clinically feasible.

Among the various treatment strategies available, the Columbus Bridge Protocol™ represents an established implant-prosthetic approach for full-arch rehabilitation through the use of implant-supported prostheses with immediate functional loading.

The non-surgical management of peri-implant diseases can be performed using a variety of tools, which are considered equivalent in effectiveness when used individually, according to the Guidelines for the Prevention and Treatment of Peri-implant Diseases. These include ultrasonic devices with implant-specific tips, titanium curettes, chitosan brushes, and air-polishing systems using glycine-based powders.

These instruments effectively remove biofilm and deposits without compromising the implant surface, unlike stainless steel curettes, which can induce microscopic alterations. Such alterations may facilitate microbial colonization and complicate effective biofilm removal.

In particular, for the removal of soft deposits, air-polishing devices with glycine powder have been shown to reduce clinical signs of inflammation in cases of peri-implant mucositis and may enhance the efficacy of non-surgical therapy in peri-implantitis. Furthermore, the use of fine-grain powders such as glycine does not cause surface alterations to the hard tissues of natural teeth or to titanium implant surfaces, nor does it lead to epithelial erosion of the soft tissues.

In patients with full-arch implant-supported prostheses, air-polishing devices represent an effective method for professional oral hygiene, including the prosthetic-mucosal interface, without requiring prosthesis removal.

Regarding home oral hygiene, the Guidelines for the Prevention and Treatment of Peri-implant Diseases do not provide universally applicable recommendations. Instead, they emphasize the importance of personalized instructions and motivation strategies, tailored to the individual needs of each patient.

For patients rehabilitated with full-arch implant-supported prostheses, in addition to compliance, prosthetic design must ensure adequate cleanability. Ideally, designs should avoid the reconstruction of soft tissues, thereby facilitating daily hygiene procedures.

The primary home-care tools recommended for these patients include manual or electric toothbrushes, sponge dental floss, and interdental brushes. The use of an angled toothbrush has also been suggested to improve access to difficult areas, such as prosthetic surfaces in direct contact with the mucosa and distal cantilevers.

ELIGIBILITY:
Inclusion Criteria:

* good general health (classified as ASA Physical Status ≤ 2, according to the American Society of Anesthesiology),
* patients with implant-supported prosthetic rehabilitation completed following the Columbus Bridge Protocol at least six months prior to enrollment

Exclusion Criteria:

* patients under the age of 18; heavy tobacco smokers (≥10 cigarettes per day);
* pregnant or breastfeeding women;
* individuals with autoimmune diseases, with or without oral tissue involvement;
* patients presenting biological complications (such as lack of osseointegration, implant mobility, or implant loss) affecting one or more implants;
* cases of peri-implantitis involving at least one implant; individuals with less than 40% peri-implant bone support as measured radiographically;
* patients taking medications known to induce gingival overgrowth, as well as those undergoing corticosteroid or antibiotic therapy in the three months prior to and during the study period, or receiving antiresorptive drug therapy;
* individuals with motor, manual, or cognitive impairments;
* patients whose full-arch implant-supported rehabilitation had been performed at other facilities;
* individuals with respiratory disorders; and those diagnosed with infectious diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Plaque on implant abutment | 3 months
  Plaque Index was recorded on the implants prior to the implementation of any procedure that could potentially lead to biofilm removal, evaluating six sites per implant. The absence or presence of plaque will be assessed using a periodontal probe

SECONDARY OUTCOMES:
Plaque on prosthesis | 3 months
  A plaque disclosing solution (Mira-2-Ton Solution, Hager & Werken GmbH & Co., Duisburg, Germany) was applied to the surfaces in contact with the mucosa, enabling the detection of residual deposits despite professional oral hygiene procedures. The biofilm was stained in shades of pink, purple, and blue.
  The prosthetic framework was analyzed using ImageJ software version 1.45s (National Institutes of Health, Bethesda, MD, USA). Following the upload of a photograph - captured with a Nikon D7500 camera equipped with a Nikon AF-S Micro NIKKOR 85 mm f/3.5G lens, with the prosthetic component placed on a flat surface covered with a green fabric and the camera positioned perpendicularly to the surface - pixels corresponding exclusively to pink, violet, and blue shades were selected, thereby isolating the plaque-stained areas. Similarly, a selection was performed to include only green pixels, corresponding to the background fabric, in order to exclude the prosthesis from the selection.
  Subsequ
Bleeding on probing on implant abutment | 3 months
  Bleeding on Probing was assessed by the presence of bleeding within 30 seconds after probing on six sites each implant.
Probing depth on implant abutment | 3 months
  Probing Depth was measured as the distance between the tip of the probe inserted into the sulcus and the margin of the peri-implant mucosa, applying an insertion force of approximately 0.2 N, at six sites per implant
Keratinized mucosa | 3 months
  Keratinized Tissue was measured as the distance between the peri-implant mucosal margin and the mucogingival junction at the buccal site of each implant.

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Città della Salute e della Scienza, Torino, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided